CLINICAL TRIAL: NCT02587416
Title: A Study of the Effect of Oral, Multiple-Dose 300 mg and 900 mg Gemcabene (CI-1027) Administration on the Steady-State Pharmacokinetics of Atorvastatin 80 mg
Brief Title: Effect of Gemcabene on the Pharmacokinetics of Atorvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A4141002
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesteremia
Keywords: Pharmacokinetics; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemcabene 300 mg (Experimental): Gemcabene 300 mg
  Interventions: Drug: Gemcabene 300 mg; Drug: Atorvastatin
- Gemcabene 900 mg (Experimental): Gemcabene 900 mg
  Interventions: Drug: Gemcabene 900 mg; Drug: Atorvastatin
- Atorvastatin 80 mg (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Gemcabene 300 mg — 1x300 mg gemcabene tablets orally once daily (QD) for 11 days
  Arms: Gemcabene 300 mg
Drug: Gemcabene 900 mg — 3x300 mg Gemcabene tablets orally once daily (QD) for 11 days
  Arms: Gemcabene 900 mg
Drug: Atorvastatin — 2x40 mg Atorvastatin tablets orally once daily (QD)

SUMMARY:
The purpose of this study is to determine the effect of gemcabene on the pharmacokinetics of atorvastatin 80 mg

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18-65 years of age
* Good health as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory measurements;
* Body weight 45 kg or greater, with a body mass index (BMI) ≤ 35 kg/m² (weight [kg]/height[meters]²)

Exclusion Criteria:

* If female, of childbearing potential or lactation
* History of significant adverse reaction to any lipid-lowering agent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2002-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | Days 5, 16 and 27
  Cmax
Pharmacokinetics | Days 5, 16, and 27
  Area Under the Curve (AUC)

SECONDARY OUTCOMES:
Adverse Events | 27 days
Clinical Laboratory - hematology, chemistry, urinalysis | 27 days
  Clinical Laboratory Abnormalities
ECG | 27 days
  Clinically Significant Changes